CLINICAL TRIAL: NCT02953028
Title: Treatment of Mild and Moderate Obstructive Sleep Apnea (OSA) by Continuous Positive Airway Pressure (CPAP) or Mandibular Advancing Splint (MAS) - a Randomized Controlled Trial on Patient Specific Factors, Success Rate and Compliance
Brief Title: Obstructive Sleep Apnea - Patient Specific Factors, Success Rate and Compliance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Tromso (Other)
Collaborators: University Hospital of North Norway (Other); Public Dental Service Competence Centre of Northern Norway (Unknown); St. Olavs Hospital (Other)
Responsible Party: Principal Investigator, Lars Martin Berg, PhD-student, University of Tromso
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSAstudie-UiT
Record Dates: First submitted 2016-02-26; First posted 2016-11-02 (Estimated); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Continuous Positive Airway Pressure; Mandibular Advancing Splint; Efficacy; Compliance; Health related quality of life; Randomized Controlled Trial; Snoring; Mandibular Advancing Appliance; Mandibular Advancing Device; Humans; Quality of Life; Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive; Patient Compliance; Snoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous Positive Airway Pressure (Active Comparator): Patients treated With an auto-CPAP-machine which is a compressor Connected to a nose- or face mask which provides increased air pressure, opening the upper Airways during an apnea or hypopnea event.
  Interventions: Device: CPAP
- Mandibular Advancing Splint (Active Comparator): Patients treated With a twin block splint (oral appliance) advancing the mandible and thereby opening the upper Airways for easier passage of air during sleep preventing apnea and hypopnea events.
  Interventions: Device: Mandibular Advancing Splint

INTERVENTIONS:
Device: CPAP — Auto-CPAP-machine for treating Obstructive Sleep Apnea With positive airway pressure
  Other Names: Resmed Autoset S9
  Arms: Continuous Positive Airway Pressure
Device: Mandibular Advancing Splint — Oral Appliance for providing an open upper airway as a mean of treating Obstructive Sleep Apnea
  Other Names: Respire Blue; Somnodent Fusion
  Arms: Mandibular Advancing Splint

SUMMARY:
Obstructive sleep apnea (OSA) is a condition where the patient's breathing cease during sleep due to collapse of the oro-pharynx. The consequences are reduced quality of sleep, increased risk for developing cardiovascular disease and increased risk of accidents caused by daytime sleepiness. Among Norwegians 30-65 yrs, the prevalence of OSA are estimated to 16%. The golden standard in OSA-treatment is Continuous Positive Airway Pressure (CPAP). This is effective and must be used for life. However, CPAP-treatment might be uncomfortable for the patient, with poor compliance as a result. An alternative is Mandibular Advancing Splints (MAS), which is perceived as less troublesome and may initiate higher compliance. Through mapping of patient characteristics, the researchers investigate which patient-type benefits most from two different treatment-devices. The aim of the study is to assess how the MAS treatment differ from the CPAP treatment in respect to efficacy, compliance and impact on health related quality of life among patient diagnosed with mild/moderate OSA. All OSA patients referred to the Ear- Nose- Throat-department (ENT) at University Hospital, Northern-Norway (UNN) and St.Olavs Hospital were invited to participate in the study. The sample size at completion of the study should be 140 patients. Participants in the trial were randomly allocated to the two treatment groups, and assessed after 4 and 12 months of treatment. Data were collected through anamnesis, clinical examination, clinical photos, radiographs and questionnaires concerning general health related quality of life (SF36), oral health, cognitive aspects (HADS), sleep quality (PSQI), daytime sleepiness (Epworth's Sleepiness scale) and compliance.

ELIGIBILITY:
Inclusion Criteria:

* 10 ≤ Apnea-Hypopnea-Index ≤ 30 at baseline
* Subjective symptoms of OSA
* Ability of at least 5mm protrusion of the mandible
* Accept randomization of treatment modality
* Accept to fill in the questionnaires
* Accept to attend at planned consultations

Exclusion Criteria:

* Primarily central sleep apnea
* Known temporomandibular dysfunction (TMD)
* Mental instability
* Drug abuse
* Extensive usage of sedative medication which disqualifies for OSA-treatment
* Extensive gag-reflex or claustrophobia
* Inadequate dental support (< 10 teeth in lower jaw)
* Inadequate periodontal support (no tooth mobility > Miller grade I)
* Anatomical abnormalities in the nasal cavity or oro-pharynx that disqualifies the use of CPAP and/or MAS
* Anatomical abnormalities which should be surgically corrected before treatment with CPAP and/or MAS
* Severely compromised general health condition
* Pregnancy
* General health issues that disqualifies the use of CPAP and or MAS

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Association between patient characteristics and adherence to treatment With either CPAP or MAS | 12 months
  Combining measurements from questionnaires at baseline and 12 months to map the patient characteristics of those patients treated for mild or moderate OSA who comply, or do not comply to CPAP-intervention or MAS-intervention respectively. Detailed description of measurements collected are listed in secondary outcome measures.

SECONDARY OUTCOMES:
Efficacy of MAS and CPAP measured by Apnea-Hypopnea-Index (AHI). Data collected by respiratory polygraphy. | 4 months
  Objective measurement of the efficacy of MAS or CPAP treatment in patients having mild or moderate OSA. Apnea-events/hypopnea-events and oxygen desaturation-index registered by respiratory polygraphy are combined to give an AHI-score before treatment and after 4 months of intervention.
Efficacy of MAS and CPAP measured by Apnea-Hypopnea-Index (AHI). Data collected by respiratory polygraphy. | 12 months
  Objective measurement of the efficacy of MAS or CPAP treatment in patients having mild or moderate OSA. Apnea-events/hypopnea-events and oxygen desaturation-index registered by respiratory polygraphy are combined to give an AHI-score before treatment and after 12 months of intervention.
Self-reported patient compliance to MAS or CPAP collected by questionnaire | 4 months
  Patient adherence to the use of MAS or CPAP in patients having mild or moderate OSA
Self-reported patient compliance to MAS or CPAP collected by questionnaire | 12 months
  Patient adherence to the use of MAS or CPAP in patients having mild or moderate OSA
Self-reported quality of life collected by the questionnaire Short Form-36 (SF-36) | 4 months
  Health related Quality of life at baseline and after 4 months of treatment with either MAS or CPAP in patients having mild or moderate OSA
Self-reported quality of life collected by the questionnaire Short Form-36 (SF-36) | 12 months
  Health related Quality of life at baseline and after 12 months of treatment with either MAS or CPAP in patients having mild or moderate OSA
Self-reported symptoms of anxiety and/or depression collected by the questionnaire Hospital Anxiety and Depression Scale (HADS) | 4 months
  Self reported signs on depression and anxiety at baseline and after 4 months of treatment with either MAS or CPAP in patients having mild or moderate OSA
Self-reported symptoms of anxiety and/or depression through the questionnaire Hospital Anxiety and Depression Scale (HADS) | 12 months
  Self reported signs on depression and anxiety at baseline and after 12 months of treatment with either MAS or CPAP in patients having mild or moderate OSA
Self-reported experience of sleep-quality through the questionnaire Pittsburgh Sleep Quality Index (PSQI) | 4 months
  Self perceived sleep quality at baseline and after 4 months of treatment with either MAS or CPAP in patients having mild or moderate OSA
Self-reported experience of sleep-quality through the questionnaire Pittsburgh Sleep Quality Index (PSQI) | 12 months
  Self perceived sleep quality at baseline and after 12 months of treatment with either MAS or CPAP in patients having mild or moderate OSA

CONTACTS AND LOCATIONS:
Overall Officials: Tordis A. Trovik, PhD, DDS, Study Chair — University of Tromsø, Department of Community Medicine
Locations (2):
- Norway (2):
  - St.Olavs Hospital, Trondheim, Sør-Trøndelag
  - University Hospital of North Norway, Tromsø, Troms

IPD SHARING:
Plan to Share IPD: No